CLINICAL TRIAL: NCT05770414
Title: Can We Still Make the Connection? Evaluating an Online Parenting Intervention for Caregivers of Infants and Young Children
Brief Title: Evaluating an Online Parenting Intervention for Caregivers of Infants and Young Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-02-23-8888
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Parent-Child Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants assigned to this group will receive the MTC online program after completing the pre-intervention questionnaire.
  Interventions: Behavioral: Make the Connection® Online Program
- Waitlist control group (No Intervention): Participants assigned to this group will not receive the MTC online program during the study period. At the end of the 8 weeks and after the post-questionnaire is completed, they will have the option to receive the MTC online program if they wish.

INTERVENTIONS:
Behavioral: Make the Connection® Online Program — Make the Connection® (MTC) is an evidence-based parenting program offered by Strong Minds Strong Kids, Psychology Canada. Recently, the MTC program has been adapted to an online platform to help increase scalability and accessibility across Canada. The online modality is self-administered by caregivers and consist of 8 weekly, 15-minute modules.
  MTC is an attachment-focused, evidence-informed, parent training program that is designed to support the development of positive parent-child relationships by teaching caregivers to understand their infant's cues. The overarching goal of the program is to enhance parental attitudes and cognitions towards their infants, which have been shown to be associated with sensitive parenting behaviour, and in turn, secure child attachment. Ultimately, by improving parenting skills and attitudes, the program seeks to support secure infant attachment.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the online modality of the Make the Connection (MTC) program in caregivers of infants and young children. The main questions it aims to answer are:

* Does the MTC online program result in changes in the child-caregiver relationship, caregiver self-competence, caregiver stress, caregiver depression, as well as caregiver and child emotion regulation, as compared to a waitlist control?
* Are caregivers who experience psychosocial risks (e.g., elevated depression scores, social isolation) deriving similar benefits in the child-caregiver relationship, caregiver self-competence, caregiver stress, caregiver depression, as well as caregiver and child emotion regulation as caregivers who are not?
* What are some of the barriers, facilitators, perceived benefits, and risks to participating in the MTC online program from the perspective of caregivers?

Participants will be randomly placed into either the intervention group or the waitlist control group. Both groups will be asked to complete a pre-intervention questionnaire, the intervention group will be invited to complete the 8-week MTC online program consisting of a weekly 15-minute module, and both groups will lastly be asked to complete a post-intervention questionnaire.

Researchers will compare the intervention group and the waitlist control group to see if the MTC online program results in improved caregiver-child bond, caregiver self-efficacy, caregiver stress, and caregiver depression.

ELIGIBILITY:
Inclusion Criteria:

* caregivers with children between the ages of 0-3 years old
* caregivers are primarily responsible for the children
* caregivers are over 18 years of age
* caregivers are able to complete the questionnaires and understand the program content in English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Caregiver-child bond will be measured using the Maternal Postnatal Attachment Scale (MPAS) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The MPAS is a 19-item questionnaire that assesses caregivers' relational attitudes towards their infant. There are three main subscales derived from the measure: Quality of Attachment, Pleasure in Interaction, and Absence of Hostility. The MPAS has shown strong psychometric properties for use in community samples and can be used with mothers and fathers. The minimum score is 19 while the maximum score is 95. Lower scores indicate more problematic responses and there is no cut off points for problematic or concerning relationships.

SECONDARY OUTCOMES:
Caregivers' self-efficacy will be measured using the Parent Sense of Competence Questionnaire (PSOC) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The PSOC has 14-items and measures a caregiver's experiences in their role as a parent. There are three substances including Interest, Efficacy, and Satisfaction. The questionnaire has been widely used to assess parenting attitudes and has adequate psychometric properties. A higher score indicates a higher parenting sense of competency. There are no average scores or 'cut-off's' for this tool.
Caregivers' stress will be measured using the Parenting Stress Scale (PSS) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The PSS is an 18-item questionnaire that assesses both positive and negative perceptions and feelings associated with being a parent. The PSS has been widely used and has been found to have strong psychometric properties. Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress. There is no cut-off score.
Caregivers' depression will be measured using the Centre for Epidemiological Studies Depression Scale (CES-D) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
  The CES-D contains 20 items and requires individuals to rate how often they experienced symptoms of depression over the past week. This scale has demonstrated good reliability and validity. Possible range of scores is 0 to 60, with higher scores indicating the presence of more symptomatology. A score of 16 or greater is considered a risk for clinical depression.
Caregivers' emotion regulation will be assessed using three items from the Difficulties in Emotion Regulation Scale (DERS) | Change from pre-intervention scores at baseline and post-intervention scores at week 8
Infant emotion regulation will be assessed using two items from the Ages & stages questionnaire: Social-Emotional, Second Edition (ASQ-SE) | Change from pre-intervention scores at baseline and post-intervention scores at week 8

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Barriault S, Deneault AA, Kempe S, Madigan S, Lovegrove A, Dimitropoulos G, Riddell RP, Racine N. A randomized waitlist control trial of the Make the Connection(R) online program for caregivers of infants and young children: Study protocol. Digit Health. 2024 Jan 9;10:20552076231221053. doi: 10.1177/20552076231221053. eCollection 2024 Jan-Dec. PMID 38205035